CLINICAL TRIAL: NCT01442909
Title: Phase IV Randomized Trial of Pemetrexed Followed by Docetaxel or in Reverse Sequence in Non-small-cell Lung Cancer Patients Failed Previous Chemotherapy
Brief Title: Pemetrexed Followed by Docetaxel or in Reverse Sequence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 97-02-09
Record Dates: First submitted 2008-05-25; First posted 2011-09-29 (Estimated); Last update posted 2011-09-29 (Estimated); Status verified 2011-09

CONDITIONS: Non-small-cell Lung Cancer
Keywords: lung cancer; docetaxel; pemetrexed
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Docetaxel; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- D followed by P (Active Comparator): Docetaxel 60 mg/m2 intravenous infusion (IV) day 1 every 3 weeks for 4-6 cycles (stable disease up to 4 cycles, partial or complete response up to 6 cycles), followed by pemetrexed 500 mg/m2 IV day 1 every 3 weeks for 4-6 cycles (stable disease up to 4 cycles, partial or complete response up to 6 cycles).
  Interventions: Drug: Docetaxel and pemetrexed
- P followed by D (Active Comparator): Pemetrexed treatment followed by docetael (in reverse sequence of Arm "D followed by P"
  Interventions: Drug: Docetaxel and pemetrexed

INTERVENTIONS:
Drug: Docetaxel and pemetrexed — docetaxel 60mg/m2 every 3 weeks for 4 cycles followed by pemetrexed 500mg/m2 every 3 weeks for 4 cycles; or in reverse sequence.
  Other Names: taxotere; alimta

SUMMARY:
Both pemetrexed and docetaxel have been reported to have similar activity against non-small cell lung cancer (NSCLC) who failed previous chemotherapy in a large randomized phase III study. However, no study showed different toxicity and efficacy profiles within individual patients. Present phase II randomized clinical trial is designed to answer these questions, with addition of information about whether or not sequential therapy can prolong disease-free and overall survival.

DETAILED DESCRIPTION:
Docetaxel was the first third-generation anti-cancer drug found to have activity in second-line chemotherapy for NSCLC, with a prolongation of patient survival in phase III randomized trials comparing docetaxel with vinorelbine or ifosfamide, or with the best supportive care, for NSCLC patients who have failed previous chemotherapy; thus, it has been recommended for the second-line treatment of NSCLC. Four years after these trials, pemetrexed showed similar activity with less toxicity, when compared with docetaxel treatment in a phase III randomized trial of NSCLC patients previously treated with chemotherapy.

Pemetrexed is a multitargeted antifolate which exhibits clinical activity in a variety of solid tumors, especially malignant mesothelioma and NSCLC. It inhibits thymidylate synthase, dihydrofolate reductase and glycinamide ribonucleotide formyl transferase. Pemetrexed has confirmed activity against previously chemotherapy-treated NSCLC and has a better toxicity profile than docetaxel, in which study docetaxel dosage used was 75 mg/m2 intravenous infusion (IV) every 3 weeks. However, docetaxel dosage used in Japan and Taiwan is usually 60 mg/m2 every 3 weeks.

Whether or not toxicity profiles of these two different drugs in same individual patients is similar to findings of patients who received specific drug only is unknown, so is unknown of toxicity profiles of docetaxel 60 mg/m2 every 3 weeks comparing alimta 500 mg/m2 every 3 weeks. Present phase II randomized clinical trial is designed to answer these questions, with addition of information about whether or not sequential therapy can prolong disease-free and overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. histologically or cytologically confirmed non-small cell bronchogenic carcinoma, inoperable stage IIIB or IV
2. aged 18 years or older
3. failed previous platinum-based chemotherapy
4. presence of at least one measurable disease which is defined as lesion that can be measured in at least 1 dimension as ≥ 20 mm with conventional CT or ≥ 10 mm with spiral CT scan
5. performance status of Eastern Cooperative Oncology Group (ECOG) 0, 1, or 2
6. white blood cell (WBC) ≥ 3,000/mm3, absolute neutrophil count (ANC) ≥ 1,500/mm3, platelets ≥ 100,000/mm3 and hemoglobin ≥ 10 mg / dl
7. serum creatinine level 2.0 mg/dL or lower
8. serum bilirubin less than 1.5 times the upper limit of normal range (ULN)
9. alanine aminotransferase (ALT) or aspartate aminotransferase (AST) less than 3 times the ULN (less than 5 times the ULN in liver metastases)
10. written informed consent to participate in the trial In addition, in female patient with childbearing potential, either terminated by surgery, radiation, or menopause, or attenuated by use of an approved contraceptive method (intrauterine contraceptive device [IUD], birth control pills, or barrier device) during and for three months after trial. Patients who previously treated by surgery are needed to demonstrate progressive disease before entering the study.

Exclusion Criteria:

1. Active infection (at the discretion of the investigator).
2. Active central nervous system (CNS) metastases.
3. Breast feeding.
4. Serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator).
5. Use of any investigational agent in the month before enrollment into the study.
6. Concomitant myelosuppressive radiotherapy to target lesion, chemotherapy, hormonal therapy, or immunotherapy will not be allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Incidence of grade III or IV leukopenia during treatment | one year

SECONDARY OUTCOMES:
progression-free survival | one year

CONTACTS AND LOCATIONS:
Overall Officials: Yuh-Min Chen, MD, PhD., Principal Investigator — Chest Department, Taipei VGH
Locations (1):
- Taipei VGH, Taipei, Taiwan